CLINICAL TRIAL: NCT00118014
Title: Sertraline and Habit Reversal in the Treatment of Patients With Trichotillomania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Michael Jenike, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1999-P-003152; 98-09272
Record Dates: First submitted 2005-07-01; First posted 2005-07-11 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Impulse Control Disorders
Keywords: Trichotillomania; Habit Reversal Training; Sertraline; Zoloft
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders; Trichotillomania | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sertraline
Behavioral: Habit Reversal Training

SUMMARY:
The purpose of this study is to assess the extent of symptom remission in patients with trichotillomania following treatment with sertraline and/or behavior therapy.

DETAILED DESCRIPTION:
The purpose of this study is to assess the extent of symptom remission in patients with trichotillomania following treatment with sertraline and/or behavior therapy.

Following entry into the study, subjects will undergo a washout period if they are currently taking a psychotropic medication (two weeks for psychotropic medications except for fluoxetine, which requires a four-week washout). Subjects will then be given a single-blind placebo for two weeks and assessed for symptom consistency.

Subjects will take sertraline or placebo in a double-blind design. Subjects will be assessed with the Hamilton Rating Scale for Depression (HAM-D-17), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Clinical Global Impressions Scale (CGI), Hair Pulling Scale (HPS), Trichotillomania (TTM) Impact Scale, Psychiatric Institute Trichotillomania Scale (PITS), National Institute of Mental Health (NIMH) Scale, and Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) at the start of the washout period and at the end of week two in order to be randomized into the study. Subject randomization to a treatment arm will be based on the random table and in equal proportions.

Subject change scores will be assessed for the above scales, and change scores for the four different treatment groups will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have a DSM-IV diagnosis of TTM.
* TTM symptoms for at least 4 months.
* Scalp as primary site of hair pulling.
* HPS score greater than or equal to 15 OR TTM Impact Scale score greater than 30.
* Written informed consent.
* Men or women aged 18-65 years old.
* Females of childbearing potential must have a negative serum beta-HCG pregnancy test.

Exclusion Criteria:

* Pregnant women or women of childbearing potential who are not using a medically accepted means of contraception.
* Patients who, in the investigator's judgement, pose a serious suicidal or homicidal risk.
* Serious or unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic disease. Patients on anticoagulant therapy.
* History of seizure disorder.
* Comorbid bipolar disorder, psychosis, organic mental disorder, or developmental disorder.
* If there is a history of substance abuse, patients must be in remission at least 6 months.
* Past trials of sertraline.
* Currently being treated with behavioral therapy, specifically habit reversal training, for TTM.
* Other medications for medical disorders that may interact with sertraline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2000-01; Primary Completion 2004-04 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions Scale change scores (week 2 versus 22) | Week 2 to 22
Hair Pulling Scale change scores (week 0 versus 22) | Week 0 to 22
TTM Impact Scale change scores (week 0 versus 22) | Week 0 to 22
PITS (week 0 versus 22) | Week 0 to 22
NIMH Scale (week 0 versus 22) | Week 0 to 22

SECONDARY OUTCOMES:
HAM-D-17 (week 0 versus 22) | Week 0 to 22
BDI (week 0 versus 22) | Week 0 to 22
BAI (week 0 versus 22) | Week 0 to 22
Q-LES-Q (week 0 versus 22) | Week 0 to 22

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jenike, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital - OCD Clinic, Charlestown, Massachusetts, United States

REFERENCES:
- [Derived] Hoffman J, Williams T, Rothbart R, Ipser JC, Fineberg N, Chamberlain SR, Stein DJ. Pharmacotherapy for trichotillomania. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD007662. doi: 10.1002/14651858.CD007662.pub3. PMID 34582562